CLINICAL TRIAL: NCT02023034
Title: EFFECTIVENESS OF VIRTUAL EXERCISES ON THE FUNCTIONAL EXERCISE CAPACITY, FATIGUE AND QUALITY OF LIFE IN PATIENTS WITH PARKINSON'S DISEASE: A RANDOMIZED CLINICAL TRIAL
Brief Title: Virtual Exercises in Patients With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade Evangelica do Parana (Other)
Responsible Party: Principal Investigator, Silvia Valderramas, Silvia Valderramas, Faculdade Evangelica do Parana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEPAR - 04
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease, Physical Therapy, Fatigue, Quality of Life
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual exercises (Experimental): All patients underwent 12 sessions, twice a week for a period of 06 weeks. The exercises were performed in the "on" dopaminergic medication, supervised by the researchers, the period instrument used was the video game with the Nintendo ® Wii Balance Board ® platform.
  Interventions: Other: Virtual exercises
- Control (Sham Comparator): Traditional exercises. All patients underwent 12 sessions, twice a week for a period of 06 weeks. The exercises were performed in the "on" dopaminergic medication, supervised by the researchers.
  Interventions: Other: Virtual exercises

INTERVENTIONS:
Other: Virtual exercises — The exercises will be performed with the Nintendo ® Wii Balance Board ® platform, and consist in: 1) Table Tilt; 2) Obstacle Course; 3) Tilt City; 4) Basic step; 5) Penguin; 6) Heading Soccer; 7) Basic Run. All patients underwent 12 sessions, twice a week for a period of 06 weeks.

SUMMARY:
Introduction: Although the motor changes are well determined in Parkinson's disease (PD), few studies describe the effects the virtual exercises on the clinical and functional outcomes in this disease.

Objectives: To analyze the effectiveness of virtual exercises on functional exercise capacity, fatigue and quality of life in patients with PD.

Methods: 20 subjects, 60 years old will be included, who will be randomized into 2 groups: group of virtual exercises associated with conventional exercises (n = 10) and control group with conventional exercise group (n = 10).

The following variables are evaluated: functional exercise through walking test in 6 minutes, fatigue by the Fatigue Severity Scale and Quality of Life through Quality of Life Questionnaire-PDQ-39.

ELIGIBILITY:
Inclusion Criteria:

* will be selected for the study
* subjects with a clinical diagnosis of Parkinson's disease
* 0-III H&Y
* 40 to 80 years
* both sexes
* with preserved cognitive stage (Mini Mental> 24).

Exclusion Criteria:

* will be excluded subjects who have some acute pain or associated diseases
* such as severe or unstable heart disease
* visual disturbances
* using some march auxiliary device, which compromise the 6MWT and exercise protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Improvement of functional exercise capacity | The subjects will be followed for a period of 90 days.
  Assessed by the 6-minute walk test (6MWT), according to the guidelines of the American Thoracic Society, which is based on the evaluation of the maximum distance traveled by the patient for six minutes, expressed in meters.

SECONDARY OUTCOMES:
Reduction of Fatigue | The subjects will be followed for a period of 90 days.
  Assessed by the Fatigue Severity Scale, which consists of a questionnaire that assesses the impact of fatigue-related activities of daily living, rating ranges from 1 to 7 where 1 indicates little tired and 7, very tired.

OTHER OUTCOMES:
Improvement of Quality of life | The subjects will be followed for a period of 90 days.
  Assessed by the specific questionnaire for Parkinson's Disease, the PDQ 39.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Valderramas, PhD, Principal Investigator — Faculdade Evangelica do Parana
Locations (1):
- Associação Paranaense dos Portadores de Parkinsonismo, Curitiba, Paraná, Brazil